CLINICAL TRIAL: NCT02102633
Title: An Open-Label, Randomized, 2-Period Crossover Study To Evaluate The Effect Of A Single Oral Dose Of Bosutinib On The Pharmacokinetics Of Dabigatran Etexilate Mesylate Administered Orally To Healthy Subjects
Brief Title: Drug Interaction Study Between Bosutinib And Dabigatran
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1871043
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: bosutinib; dabigatran; drug interaction; p-glycoprotein; pharmacokinetics
MeSH Terms: interventions — Dabigatran; bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dabigatran (Experimental): Dabigatran 150 mg orally
  Interventions: Drug: Dabigatran
- Dabigatran + Bosutinib (Experimental): Dabigatran 150 mg co-administered with Bosutinib 500 mg orally
  Interventions: Drug: Bosutinib; Drug: Dabigatran

INTERVENTIONS:
Drug: Dabigatran — Dabigatran 150 mg orally
  Arms: Dabigatran
Drug: Bosutinib — Bosutinib 500 mg orally
  Arms: Dabigatran + Bosutinib
Drug: Dabigatran — Dabigatran 150 mg orally
  Arms: Dabigatran + Bosutinib

SUMMARY:
The study evaluates the effect of a single oral dose of bosutinib on the single dose pharmacokinetics of dabigatran, a p-glycoprotein substrate, in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between 21 to 55 years old and BMI between 17.5 and 30.5 kg/m2.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Risks of bleeding including prior personal or familiar history of abnormal bleeding, hereditary or acquired coagulation or platelet disorder or abnormal coagulation test (PT/INR or PTT/aPTT greater than upper limit of normal) result at screening.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of non-hormonal contraception as outlined in this protocol from at least 14 days prior to the first dose of study medication.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 48 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Maximum Observed Plasma Concentration (Cmax) | 48 hours
  Maximum Observed Plasma Concentration

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 48 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 48 hours
  Time to Reach Maximum Observed Plasma Concentration
Plasma Decay Half-Life (t1/2) | 48 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | 48 hours
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 48 hours
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, DeLand, Florida, United States

REFERENCES:
- [Derived] Hsyu PH, Pignataro DS, Matschke K. Effect of bosutinib on the absorption of dabigatran etexilate mesylate, a P-glycoprotein substrate, in healthy subjects. Eur J Clin Pharmacol. 2017 Jan;73(1):57-63. doi: 10.1007/s00228-016-2115-0. Epub 2016 Oct 7. PMID 27717999
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1871043&StudyName=Drug%20Interaction%20Study%20Between%20Bosutinib%20And%20Dabigatran